CLINICAL TRIAL: NCT05046899
Title: A Prospective, Randomized, Intra-patient Investigation to Assess the Clinical Performance and Safety of BIOpH+ Psoriasis Medical Bath for 8 Weeks of Treatment in Subjects With Mild to Moderate Plaque Psoriasis of Affected Body Area.
Brief Title: Investigation With BiopH+Psoriasis Medical Bath in Subject With Mild to Moderate Plaque Psoriasis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biocool AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BioC002
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Intervention Model Description: Intra-patient design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIOpH+ Psoriasis Medical Bath (Experimental): BIOpH+ Psoriasis Medical Bath is bath. Each bath will take 20 minutes and number of bath during the entire study period is approximately 35 baths.
  Interventions: Device: BIOpH+ Psoriasis Medical Bath
- Comparative device (Active Comparator): Comparative device is Cetaphil Moisturizing Lotion. The lotion will be applied on the affected body area on the same days as the BIOpH+ Psoriasis Medical Bath is performed.
  Interventions: Device: Cetaphil Moisturizing Lotion

INTERVENTIONS:
Device: BIOpH+ Psoriasis Medical Bath — 20 min bath every day during 1 week and thereafter 20 min bath every second day for additional 7 weeks.
  Arms: BIOpH+ Psoriasis Medical Bath
Device: Cetaphil Moisturizing Lotion — Cetaphil Moisturizing Lotion will be applied on the affected body area on the same days as the BIOpH+ Psoriasis Medical Bath is performed.
  Arms: Comparative device

SUMMARY:
The purpose of this investigation is to assess performance and safety of BIOpH+ Psoriasis Medical Bath in comparison to a comparative device.

DETAILED DESCRIPTION:
After being informed about the investigation and the potential risks, all subjects giving written informed consent will undergo screening to determine eligibility for study entry. At week 0, subjects who meet the eligibility requirements will be randomised in open, intra-patient investigation, treated with BIOpH+ Psoriasis Medical Bath on one side, and comparative treatment on the other side for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreed to participation and has duly signed Informed Consent Form
* Males and females ≥ 18 years of age
* In the Investigator's opinion, the patient is not likely to become pregnant during study participation (e.g. in a same-sex relationship, not sexually active, sterile, not of child-bearing age, uses contraception, etc.)
* Subject diagnosed with stable mild-moderate plaque psoriasis, defined by PASI ≤ 9
* Intra-individual difference between left and right hemi-body PASI scores not > 1.0
* Patients with symmetrical psoriasis

Exclusion Criteria:

* Presence of other forms of psoriasis other than psoriasis vulgaris (palmoplantar psoriasis, inverse psoriasis, other forms of hyperkeratosis)
* Use of systemic/biological treatment for psoriasis
* Known hypersensitivity or allergy to study products
* Any serious medical condition that could interfere with the evaluation of study results
* Poor compliance in other investigational study, as assessed by investigator
* Pregnant, breastfeeding, or planning to become pregnant during study
* Patients with alcohol -or drug abuse
* Any other conditions as judged by the investigator may make the follow-up or investigation inappropriate
* Anyone unsuitable to participate as subject according to the Declaration of Helsinki

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Change in Psoriasis Area and Severity Index (PASI) score from Baseline compared to week 8. | Baseline and week 8.
  The PASI score is a validated, investigator instrument assessing the severity of psoriasis. The severity is combined with the percentage of affected area.

SECONDARY OUTCOMES:
Dermatology Life Quality Index (DLQI) | Baseline and week 8.
  A quality of life instrument and will evaluate how much the skin problems affects the study subject's daily life. It is a 10-question questionnaire. Each question contains four response categories: 0=not at all, 1=a little, 2=a lot, and 3=very much. A higher score means worse outcome.
Psoriasis Area Severity Index (PASI) | Week 2 and week 4
  It combines the severity (erythema, induration and desquamation) and percentage of affected area. A high score means worse outcome.
  The body is divided into 4 sections:
  1. Head, weight = 0.1
  2. Arms, weight = 0.2
  3. Trunk, weight = 0.3
  4. Legs, weight = 0.4
  For each section, the percent of area of skin involved is estimated and graded:
  0. 0% of involved area
  1. <10% of involved area
  2. 10-29% of involved area
  3. 30-49% of involved area
  4. 50-69% of involved area
  5. 70-89% of involved area
  6. 90-100% of involved area Within each area, the severity is estimated for 3 clinical signs: erythema (redness), induration (thickness) and desquamation (scaling). Severity is measured on a scale from 0-4, from none to maximum.
  The sum of all 3 severity parameters is calculated for each body section, multiplied by the area score for that area, and multiplied for the weight of the body section, for a maximum score of 72.
Physician Global Assessment (PGA) | Baseline, week 2, 4, and 8
  The Physician Global Assessment, is a 5-point scoring system that will be used to assess the overall disease severity. This treatment response on each visit will be scored: 0 =cleared, 1=almost clear, 2=mild 3=moderate, and 4=severe. A higher scores mean worse outcome.
Tolerability assessment | Week 2, 4 and week 8.
  Tolerability assessment completed by the study subject about local tolerance regarding experience of pruritus and burning/stinging measured on a 5-point scale, or by questions to be answered with yes or no.
Usability /satisfaction assessments | Week 8
  A questionnaire to be answered by study subject about investigational device usability and satisfaction measured on a 5-point scale, or by questions to be answered with yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lundvall, MD, Principal Investigator — Research Unit, University Hospital Örebro, Sweden
Locations (1):
- Avdelningen för klinisk prövning, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No